CLINICAL TRIAL: NCT01156792
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Five-Treatment, Four 6-Week Period Cross-Over, Multi-Center Study to Evaluate the Effect of Adding GSK2190915 100mg, GSK2190915 300mg, Montelukast 10mg or Placebo Tablets Once Daily or Salmeterol 50mcg Inhalation Powder Twice Daily to Fluticasone Propionate 100mcg Inhalation Powder Twice Daily in Uncontrolled Asthmatic Subjects ≥ 12 Years of Age
Brief Title: Safety and Efficacy Study of Adding GSK2190915 to Low Dose Inhaled Corticosteroid Treatment for Asthma Subjects > or = 12 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114255
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: asthma; GSK2190915
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- FP 100mcg BID plus GSK2190915 100mg QD (AM) (Experimental): FP 100mcg BID plus GSK2190915 100mg QD (AM)
  Interventions: Drug: FP 100; Drug: GSK2190915 100
- FP 100mcg BID plus GSK2190915 300mg QD (AM) (Experimental): FP 100mcg BID plus GSK2190915 300mg QD (AM)
  Interventions: Drug: FP 100; Drug: GSK2190915 300
- FP 100mcg BID plus montelukast 10mg QD (PM) (Active Comparator): FP 100mcg BID plus montelukast 10mg QD (PM)
  Interventions: Drug: FP 100; Drug: montelukast
- FP 100mcg BID plus placebo BID (Active Comparator): FP 100mcg BID plus placebo BID
  Interventions: Drug: FP 100; Drug: placebo
- FP/SAL 100/50mcg BID plus placebo BID (Active Comparator): FP/SAL 100/50mcg BID plus placebo BID
  Interventions: Drug: placebo; Drug: FP/SAL 100/50

INTERVENTIONS:
Drug: FP 100 — FP 100mcg BID
  Arms: FP 100mcg BID plus GSK2190915 100mg QD (AM); FP 100mcg BID plus GSK2190915 300mg QD (AM); FP 100mcg BID plus montelukast 10mg QD (PM); FP 100mcg BID plus placebo BID
Drug: GSK2190915 100 — GSK2190915 100mg QD (AM)
  Arms: FP 100mcg BID plus GSK2190915 100mg QD (AM)
Drug: GSK2190915 300 — GSK2190915 300mg QD (AM)
  Arms: FP 100mcg BID plus GSK2190915 300mg QD (AM)
Drug: montelukast — montelukast 10mg QD (PM)
  Arms: FP 100mcg BID plus montelukast 10mg QD (PM)
Drug: placebo — placebo BID
  Arms: FP 100mcg BID plus placebo BID; FP/SAL 100/50mcg BID plus placebo BID
Drug: FP/SAL 100/50 — FP/SAL 100/50mcg BID
  Arms: FP/SAL 100/50mcg BID plus placebo BID

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of adding GSK2190915 100mg, GSK2190915 300mg or placebo tablets administered once daily to fluticasone propionate 100mcg inhalation administered twice daily in uncontrolled asthmatic subjects > or = 12 years of age over the course of 6 weeks treatment.

The secondary objectives are to undertake an exploratory analysis of the efficacy and safety of adding montelukast 10mg administered once daily or salmeterol 50mcg administered twice daily to fluticasone propionate 100mcg inhalation administered twice daily and to investigate the pharmacokinetics and pharmacodynamics of GSK2190915 in uncontrolled asthmatic subjects > or = 12 years of age over the course of 6 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 years of age or older
* Non-, former or current smokers with a documented smoking history of ≤ 10 pack years
* Asthma diagnosis as defined by the National Institutes of Health
* Best FEV1 of 50% to <80% of the predicted normal value
* Post-albuterol FEV1/FVC ratio of >0.70 at Visit 1/1a (between 5:00AM and 12:00 noon)
* ≥ 12% and ≥200mL reversibility of FEV1
* Must have been using FP 100mcg inhalation powder BID for at least 2 weeks just prior to Visit 1.
* Must be able to replace their current short-acting beta2-agonists with albuterol inhalation aerosol
* Must be able and willing to give written informed consent to take part in the study.
* Must be able and willing to comply with all aspects of the study including completion of daily e-Diary.

Exclusion criteria:

* History of life-threatening asthma
* Recent asthma exacerbation
* Concurrent respiratory disease
* Recent respiratory infection
* Liver disease
* Other concurrent diseases/abnormalities
* Oral candidiasis
* Drug allergy
* Milk protein allergy
* Immunosuppressive Medications
* Administration of systemic, oral or depot corticosteroids within 12 weeks of Visit 1
* OATP1B1 substrates within 4 weeks of Visit 1
* Cytochrome P450 3A4 (CYP 3A4) Inhibitors
* Cytochrome P450 3A4 (CYP 3A4) Inducers
* Investigational Medications
* Compliance: any infirmity, disability, or geographical location which seems likely (in the opinion of the Investigator) to impair compliance with any aspect of this study protocol
* Affiliation with Investigator's Site

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (31):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Snowise NG, Clements D, Ho SY, Follows RM. Addition of a 5-lipoxygenase-activating protein inhibitor to an inhaled corticosteroid (ICS) or an ICS/long-acting beta-2-agonist combination in subjects with asthma. Curr Med Res Opin. 2013 Dec;29(12):1663-74. doi: 10.1185/03007995.2013.842163. Epub 2013 Sep 19. PMID 24010736
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114255 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 341 participants (par.) were screened, and 162 participants were randomized. A protocol amendment necessitated withdrawal of all male participants and further enrollment of female participants only.
Pre-assignment Details: Par. meeting screening criteria, self-administered open-label fluticasone propionate 100 micrograms (µg) twice daily for 14-28 days. Eligible par. were assigned to 1 of 10 treatment sequences, receiving 4 of 5 double-blind treatments. Par. aged 12-14 years did not receive montelukast. Rescue medication (albuterol inhalation) was provided.
Groups:
- All Treatments Combined: In a total of 4 treatment periods (each of 6 weeks - the first 3 weeks considered as active washout), participants received 4 of the 5 possible treatments (A/B/C/D/E) in a double-blind double-dummy, cross-over manner. Fluticasone propionate (FP) 100 µg oral inhalation was a part of each treatment. Added regimen were, A: GSK2190915 100 milligrams (mg) once daily (OD), B: GSK2190915 300 mg OD, C: montelukast 10 mg OD, D: placebo twice daily (BID), E: salmeterol 50 µg and placebo BID. Albuterol aerosol was provided as a rescue inhalation.
Period: Overall Study
Arm/Group | All Treatments Combined
Started | 162
Completed | 93
Not Completed | 69
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 36
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 9
Not completed — other Sponsor Decision (Protocol Amendme | 11

BASELINE CHARACTERISTICS:
Arm/Group | All Treatments Combined
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 42
  American Indian or Alaska Native | 1
  Asian - Central/South Asian Heritage | 1
  White - White/Caucasian/European Heritage | 115
  Mixed Race | 2
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Trough (AM Pre-dose and Pre-rescue Bronchodilator) Forced Expiratory Volume in 1 Second (FEV1) at the End of the 6-week Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured electronically using spirometry, prior to study medication and any rescue albuterol (bronchodilator) use. At the end of the 6-week treatment period, FEV1 was measured approximately 24 hours after the participant's last morning dose of study medication and approximately 12 hours after the evening dose of study medication. Trough FEV1 was analyzed using mixed effect analysis of covariance (ANCOVA) model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effect of participant. Intent-to-Treat Population is defined as all participants who were randomized and received at least one dose of study drug.
Time Frame: End of Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Groups:
- FP + Placebo: Participants received FP 100 µg oral inhalation twice daily (BID) for 6 weeks (first 3 weeks considered as active washout), in one of the 4 treatment periods. Placebo administered every morning (AM) was added to the dosing regimen. Blinding was maintained by administration of a montelukast-matching placebo capsule every evening (PM). Albuterol aerosol was provided as a rescue inhalation.
- FP + GSK2190915 100 mg: Participants received FP 100 µg oral inhalation BID for 6 weeks (first 3 weeks considered as active washout), in one of the 4 treatment periods. GSK2190915 100 mg AM was added to the dosing regimen. Blinding was maintained by PM administration of a montelukast-matching placebo capsule. Albuterol aerosol was provided as a rescue inhalation.
- FP + GSK2190915 300 mg: Participants received FP 100 µg oral inhalation BID for 6 weeks (first 3 weeks considered as active washout), in one of the 4 treatment periods. GSK2190915 300 mg AM was added to the dosing regimen. Blinding was maintained by PM administration of a montelukast-matching placebo capsule. Albuterol aerosol was provided as a rescue inhalation.
- FP + Montelukast: Participants received FP 100 µg oral inhalation BID for 6 weeks (first 3 weeks considered as active washout), in one of the 4 treatment periods. Montelukast 10 mg capsule administered PM was added to the dosing regimen. Blinding was maintained by AM administration of GSK2190915-matching placebo tablets. Albuterol aerosol was provided as a rescue inhalation.
- FP / Salmeterol: Participants received a combination of FP 100 µg and salmeterol 50 µg oral inhalation BID for 6 weeks (first 3 weeks considered as active washout), in one of the 4 treatment periods. Montelukast 10 mg capsule administered PM was added to the dosing regimen. Blinding was maintained by AM administration of GSK2190915-matching placebo tablets and PM administration of a montelukast-matching placebo capsule. Albuterol aerosol was provided as a rescue inhalation.
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 93 | 94 | 93
Liters (L) | 2.36 (0.03) | 2.39 (0.03) | 2.40 (0.03) | 2.42 (0.03) | 2.43 (0.03)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.02 to 0.07]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.00 to 0.09]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [0.01 to 0.10]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = 0.074, 95% CI 2-sided [0.03 to 0.12]

2. Secondary Outcome: Daily Trough (Morning Pre-dose and Pre-rescue Bronchodilator) Morning Peak Expiratory Flow (PEF) Averaged Over the Last 3 Weeks of the 6-week Treatment Period
Description: The PEF is a measure of lung function and measures how fast a person can breathe out. Trough PEF was measured every morning prior to study medication dose and any rescue albuterol (bronchodilator) use. Participants recorded PEF in a daily electronic diary (eDiary). Daily trough morning PEF was averaged over the last 3 weeks of the 6-week treatment period, and analyzed using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
Liters/minute (L/min) | 349.19 (4.08) | 350.14 (4.06) | 354.96 (4.07) | 354.17 (4.05) | 361.33 (4.05)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.751, Mixed Models Analysis; Mean Difference (Final Values) = 0.946, 95% CI 2-sided [-4.91 to 6.81]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.049, Mixed Models Analysis; Mean Difference (Final Values) = 5.771, 95% CI 2-sided [0.03 to 11.51]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.123, Mixed Models Analysis; Mean Difference (Final Values) = 4.983, 95% CI 2-sided [-1.35 to 11.32]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 12.140, 95% CI 2-sided [5.93 to 18.35]

3. Secondary Outcome: Daily Evening PEF Averaged Over the Last 3 Weeks of the 6-week Treatment Period
Description: The PEF is a measure of lung function and measures how fast a person can breathe out. PEF was measured every evening prior to study medication dose and any rescue albuterol (bronchodilator) use. Participants recorded PEF in a daily eDiary. Daily evening PEF was averaged over the last 3 weeks of the 6-week treatment period, and analyzed using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
L/min | 354.06 (4.03) | 355.71 (4.02) | 359.16 (4.03) | 358.88 (4.01) | 364.35 (4.00)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.563, Mixed Models Analysis; Mean Difference (Final Values) = 1.651, 95% CI 2-sided [-3.97 to 7.27]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.072, Mixed Models Analysis; Mean Difference (Final Values) = 5.100, 95% CI 2-sided [-0.47 to 10.67]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis; Mean Difference (Final Values) = 4.822, 95% CI 2-sided [-1.37 to 11.02]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 10.292, 95% CI 2-sided [4.21 to 16.38]

4. Secondary Outcome: Daily (Average of Morning and Evening) PEF Averaged Over the Last 3 Weeks of the 6 -Week Treatment Period Between GSK2190915 and Montelukast Groups
Description: The PEF is a measure of lung function and measures how fast a person can breathe out. PEF was measured every morning and evening prior to study medication dose and any rescue albuterol (bronchodilator) use. Participants recorded PEF in a daily eDiary. Daily average of morning and evening PEF was averaged over the last 3 weeks of the 6-week treatment period, and analyzed using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant. This outcome measure explored the efficacy between GSK2190915 and montelukast due to the dosing time difference.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast
Number analyzed (Participants) | 93 | 92 | 93
L/min | 352.37 (3.90) | 356.16 (3.91) | 356.52 (3.90)
Statistical Analysis 1: Comparison: FP + GSK2190915 100 mg vs FP + Montelukast; Test type: Superiority or Other; Mean Difference (Final Values) = -4.154, 95% CI 2-sided [-9.36 to 1.06]
Statistical Analysis 2: Comparison: FP + GSK2190915 300 mg vs FP + Montelukast; Test type: Superiority or Other; Mean Difference (Final Values) = -0.364, 95% CI 2-sided [-6.22 to 5.50]

5. Secondary Outcome: Daily Asthma Symptom Score Averaged Over the Last 3 Weeks of the 6-week Treatment Period
Description: Daytime and night time asthma symptoms were recorded every evening at bedtime and every morning upon rising, respectively, before taking any rescue or study medication and before assessing the PEF. Symptoms were recorded on scales ranging from '0' (implying no symptoms) to either 5 (for daytime symptoms) or 4 (for night time symptoms) (implying severe symptoms). Participants recorded the symptoms in a daily eDiary. 24-hour period asthma symptom scores were averaged over the last 3 weeks of the 6-week treatment period, and analyzed using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 90 | 92 | 93 | 95
Score on a scale | 2.26 (0.12) | 2.26 (0.12) | 2.15 (0.12) | 2.22 (0.12) | 2.25 (0.12)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.957, Mixed Models Analysis; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.18 to 0.17]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.213, Mixed Models Analysis; Mean Difference (Final Values) = -0.108, 95% CI 2-sided [-0.28 to 0.06]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.647, Mixed Models Analysis; Mean Difference (Final Values) = -0.038, 95% CI 2-sided [-0.20 to 0.12]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.894, Mixed Models Analysis; Mean Difference (Final Values) = -0.011, 95% CI 2-sided [-0.17 to 0.15]

6. Secondary Outcome: Daily Rescue Short-acting beta2-agonist (SABA) Use Averaged Over the Last 3 Weeks of the 6-week Treatment Period
Description: A SABA (albuterol) was provided to participants as a rescue medication, to use as needed for symptomatic relief of asthma symptoms. Participants were required to record their albuterol use in the morning and in the evening. Participants recorded the number of inhalations of rescue medication in a daily eDiary. The daily rescue SABA use was averaged over the last 3 weeks of the 6-week treatment period, and analyzed using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Number of inhalations
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 90 | 92 | 93 | 95
Number of inhalations | 2.17 (0.13) | 2.14 (0.13) | 2.03 (0.13) | 2.09 (0.13) | 2.08 (0.13)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.811, Mixed Models Analysis; Mean Difference (Final Values) = -0.025, 95% CI 2-sided [-0.23 to 0.18]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.200, Mixed Models Analysis; Mean Difference (Final Values) = -0.133, 95% CI 2-sided [-0.34 to 0.07]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.415, Mixed Models Analysis; Mean Difference (Final Values) = -0.076, 95% CI 2-sided [-0.26 to 0.11]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.358, Mixed Models Analysis; Mean Difference (Final Values) = -0.084, 95% CI 2-sided [-0.26 to 0.10]

7. Secondary Outcome: Percentage of Symptom-free Days During the Last 3 Weeks of the 6-week Treatment Period
Description: Daytime asthma symptoms were recorded every evening at bedtime, before taking any rescue or study medication and before assessing the PEF. Symptoms were recorded on a 6-point scale ranging from '0' (implying no symptoms) to 5 (implying severe symptoms). Participants recorded the symptoms in a daily eDiary. The number of days when symptoms were not experienced ("symptom-free days") during the last 3 weeks of the 6-week treatment period were counted, and percentage calculated by dividing by 21 and multiplying by 100. Analysis was done using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
Percentage of days | 30.84 (3.04) | 33.51 (3.02) | 36.14 (3.03) | 34.88 (3.01) | 35.45 (3.02)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.285, Mixed Models Analysis; Mean Difference (Final Values) = 2.666, 95% CI 2-sided [-2.24 to 7.57]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis; Mean Difference (Final Values) = 5.300, 95% CI 2-sided [0.38 to 10.22]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis; Mean Difference (Final Values) = 4.036, 95% CI 2-sided [-0.63 to 8.70]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.047, Mixed Models Analysis; Mean Difference (Final Values) = 4.602, 95% CI 2-sided [0.06 to 9.14]

8. Secondary Outcome: Percentage of Symptom-free Nights During the Last 3 Weeks of the 6 Week Treatment Period
Description: Night time asthma symptoms were recorded every morning upon rising, before taking any rescue or study medication and before assessing the PEF. Symptoms were recorded on a 5-point scale ranging from '0' (implying no symptoms) to 4 (implying severe symptoms). Participants recorded the symptoms in a daily eDiary. The number of nights when symptoms were not experienced ("symptom-free nights") during the last 3 weeks of the 6-week treatment period were counted, and percentage calculated by dividing by 21 and multiplying by 100. Analysis was done using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
Percentage of nights | 37.21 (2.87) | 38.22 (2.85) | 40.55 (2.85) | 37.70 (2.84) | 38.47 (2.85)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis; Mean Difference (Final Values) = 1.014, 95% CI 2-sided [-3.64 to 5.67]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.156, Mixed Models Analysis; Mean Difference (Final Values) = 3.349, 95% CI 2-sided [-1.29 to 7.98]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.822, Mixed Models Analysis; Mean Difference (Final Values) = 0.496, 95% CI 2-sided [-3.83 to 4.82]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.555, Mixed Models Analysis; Mean Difference (Final Values) = 1.260, 95% CI 2-sided [-2.94 to 5.46]

9. Secondary Outcome: Percentage of Rescue-free Days During the Last 3 Weeks of the 6-week Treatment Period
Description: Albuterol was provided as a rescue medication, and participants were required to record rescue medication use in the morning and in the evening. Participants recorded the number of inhalations of rescue medication in a daily eDiary. The number of days when rescue medication was not used ("rescue-free days") during the last 3 weeks of the 6-week treatment period were counted, and percentage calculated by dividing by 21 and multiplying by 100. Analysis was done using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
Percentage of days | 40.44 (3.05) | 42.43 (3.03) | 42.59 (3.04) | 42.77 (3.02) | 41.96 (3.03)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.367, Mixed Models Analysis; Mean Difference (Final Values) = 1.992, 95% CI 2-sided [-2.35 to 6.33]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.332, Mixed Models Analysis; Mean Difference (Final Values) = 2.147, 95% CI 2-sided [-2.20 to 6.49]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.277, Mixed Models Analysis; Mean Difference (Final Values) = 2.331, 95% CI 2-sided [-1.88 to 6.55]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.467, Mixed Models Analysis; Mean Difference (Final Values) = 1.521, 95% CI 2-sided [-2.59 to 5.63]

10. Secondary Outcome: Percentage of Rescue-free Nights During the Last 3 Weeks of the 6-week Treatment Period
Description: Albuterol was provided as a rescue medication, and participants were required to record rescue medication use in the morning and in the evening. Participants recorded the number of inhalations of rescue medication in a daily eDiary. The number of nights when rescue medication was not used ("rescue-free nights") during the last 3 weeks of the 6-week treatment period were counted, and percentage calculated by dividing by 21 and multiplying by 100. Analysis was done using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
Percentage of nights | 45.12 (2.87) | 45.69 (2.85) | 48.79 (2.86) | 45.32 (2.85) | 43.98 (2.85)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.789, Mixed Models Analysis; Mean Difference (Final Values) = 0.575, 95% CI 2-sided [-3.65 to 4.80]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.087, Mixed Models Analysis; Mean Difference (Final Values) = 3.669, 95% CI 2-sided [-0.54 to 7.87]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.923, Mixed Models Analysis; Mean Difference (Final Values) = 0.200, 95% CI 2-sided [-3.84 to 4.24]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis; Mean Difference (Final Values) = -1.137, 95% CI 2-sided [-5.08 to 2.81]

11. Secondary Outcome: Percentage of Nights Without Awakenings Due to Asthma During the Last 3 Weeks of the 6-week Treatment Period
Description: Night time asthma symptoms were recorded every morning upon rising, before taking any rescue or study medication and before assessing the PEF. Symptoms were recorded on a 5-point scale: 0 = no symptoms during the night, 1 = symptoms causing to wake once, 2 = symptoms causing to wake twice or more, 3 = symptoms causing to be awake most of the night, 4 = could not sleep due to severe symptoms. Participants recorded the symptoms in a daily eDiary. The number of nights with no awakenings due to asthma during the last 3 weeks of the 6-week treatment period were counted, and percentage calculated by dividing by 21 and multiplying by 100. Analysis was done using mixed effect ANCOVA model for treatment effects, incorporating fixed effects of baseline, period, age, center, smoking status, and random effects of participant.
Time Frame: Week 4 to Week 6
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 92 | 92 | 92 | 93 | 95
Percentage of nights | 37.21 (2.87) | 38.22 (2.85) | 40.55 (2.85) | 37.70 (2.84) | 38.47 (2.85)
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis; Mean Difference (Final Values) = 1.014, 95% CI 2-sided [-3.64 to 5.67]
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.156, Mixed Models Analysis; Mean Difference (Final Values) = 3.349, 95% CI 2-sided [-1.29 to 7.98]
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.822, Mixed Models Analysis; Mean Difference (Final Values) = 0.496, 95% CI 2-sided [-3.83 to 4.82]
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.555, Mixed Models Analysis; Mean Difference (Final Values) = 1.260, 95% CI 2-sided [-2.94 to 5.46]

12. Secondary Outcome: Number of Participants Withdrawn Due to Lack of Efficacy During the Last 3 Weeks of the 6-week Treatment Period
Description: Participants were withdrawn if they met any of the following three criteria for 'lack of efficacy': 1) Clinic FEV1 below the FEV1 'Stability Limit' value, 2) During any consecutive 7-day period, the participant experienced PEF fallen below the PEF 'Stability Limit' for more than 3 days, or if >= 12 inhalations per day of albuterol were used for more than 2 days, and 3) Ashtma exacerbation. The number of withdrawals due to lack of efficacy were summarized for each treatment and Fisher's Exact test was used for comparison with placebo add-on. Withdrawals occurring during active washout periods are not included.
Time Frame: Week 4 to Week 6
Population: ITT Population.
Measure: Number; unit: Number of participants
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Number analyzed (Participants) | 104 | 103 | 96 | 99 | 104
Number of participants | 9 | 5 | 3 | 7 | 5
Statistical Analysis 1: Comparison: FP + Placebo vs FP + GSK2190915 100 mg; Test type: Superiority or Other; p = 0.408, Fisher Exact
Statistical Analysis 2: Comparison: FP + Placebo vs FP + GSK2190915 300 mg; Test type: Superiority or Other; p = 0.138, Fisher Exact
Statistical Analysis 3: Comparison: FP + Placebo vs FP + Montelukast; Test type: Superiority or Other; p = 0.797, Fisher Exact
Statistical Analysis 4: Comparison: FP + Placebo vs FP / Salmeterol; Test type: Superiority or Other; p = 0.408, Fisher Exact

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AE) and serious adverse events (SAE) were collected from the start of treatment until the follow-up contact (a maximum of 178 days).
Description: On-treatment AEs and SAEs are reported for the ITT Population.
Arm/Group | FP + Placebo | FP + GSK2190915 100 mg | FP + GSK2190915 300 mg | FP + Montelukast | FP / Salmeterol
Serious Adverse Events (participants affected / at risk) | 0/104 | 1/103 | 0/96 | 0/99 | 0/104
Other Adverse Events (participants affected / at risk) | 8/104 | 3/103 | 4/96 | 1/99 | 1/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FP + Placebo (N=104) | FP + GSK2190915 100 mg (N=103) | FP + GSK2190915 300 mg (N=96) | FP + Montelukast (N=99) | FP / Salmeterol (N=104)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FP + Placebo (N=104) | FP + GSK2190915 100 mg (N=103) | FP + GSK2190915 300 mg (N=96) | FP + Montelukast (N=99) | FP / Salmeterol (N=104)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1 | 1 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.